CLINICAL TRIAL: NCT01794767
Title: Normal Saline Versus Heparinized Solution Flush for Maintaining Patency of Peripheral Venous Catheters in Children
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: difficult recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Filippo Festini, Professor of Nursing, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Heparin2012
Record Dates: First submitted 2013-01-29; First posted 2013-02-20 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Infection of Intravenous Catheter; Phlebitis; Extravasation of Diagnostic and Therapeutic Materials
Keywords: peripheral venous catheter, children.
MeSH Terms: conditions — Phlebitis; Extravasation of Diagnostic and Therapeutic Materials | interventions — Saline Solution; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0,9% NaCl flush (Active Comparator): for children enrolled in this group, the nurse will perform the flushing of peripheral venous catheter using flush-solution as a bolus with saline 0.9% NaCl in the amount (ml) needed to fill the entire circuit of the catheter. The flushing will be performed routinely at the end of each fleboclisis
  Interventions: Drug: 0,9% NaCl flush
- Heparin 50U/ml (Experimental): for children enrolled in this group, the nurse will perform the washing of peripheral venous catheter using flush-solution as a bolus with heparin 50U/ml in the amount (ml) needed to fill the entire circuit of the catheter. The washing will be performed routinely at the end of each fleboclis
  Interventions: Drug: Heparin 50U/ml

INTERVENTIONS:
Drug: 0,9% NaCl flush — Normal Saline solution
  Other Names: Normal Saline
  Arms: 0,9% NaCl flush
Drug: Heparin 50U/ml — Heparin solution
  Other Names: Heparin solution 50 U/ml, Epsodilave
  Arms: Heparin 50U/ml

SUMMARY:
The aim of the study is to verify if the periodic flush with normal saline 0.9% NaCl causes a longer or equal duration of patency of peripheral venous catheters, compared with heparin solution 50 U / ml flush, in children from 2 years to 14 years. Only 22 and 24 gauge catheters Will be included in the study.The study will assess in particular:

* the difference of permanence in situ of the device
* the difference in incidence of complications (in detail: obstruction, phlebitis, thrombocytopenia, systemic anticoagulation)
* the difference in costs between use of saline normal saline 0.9% NaCl solution and heparinized 50 U / ml.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 years and 14 years old
* Medical prescription of intravenous antibiotic therapy for at least 2 doses on the day
* Presence of informed consent to participate to the study provided by the parents
* No known hypersensitivity to heparin
* No known hypersensitivity to the patch fixing materials (polyurethane and / or glue)
* Absence of diseases buoyancy coagulation (haemophilias and / or thrombophilias)
* No antecedents trombopenie dued to the use of any type of heparin or a pentosan polysulfate
* No existing treatment based on corticosteroids and / or anti-inflammatory

Exclusion Criteria:

* age outside the range 2 - 14 years
* children for which there is no prescription of intravenous antibiotic therapy for at least 2 times a day
* children for which the parents have not consented to the study
* children with known hypersensitivity to heparin
* children with known hypersensitivity to the patch fixing materials (polyurethane and / or adhesive)
* children with disease-causing buoyancy coagulation (Hemophilia and / or thrombophilia)
* children with antecedents of trombopenie occurring by the use of any type of heparin or of a pentosan polyphosphate
* children in treatment with corticosteroids and / or anti-inflammatory

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Average length of stay on site of the catheter measured in hours | participants will be followed for the duration on site of the first peripheral venous catheter inserted to each recruited subject, i.e. for an expected average of 10 dayse

SECONDARY OUTCOMES:
Incidence of complications extimated overall and by type of complication | participants will be followed for the duration on site of the first peripheral venous catheter inserted to each recruited subject, i.e. for an expected average of 10 days
Average cost for the maintenance of the catheter of each subject (pro day and in total) | participants will be followed for the duration on site of the first peripheral venous catheter inserted to each recruited subject, i.e. for an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Festini, RN, BSN, MSN, Principal Investigator — University of Florence
Locations (1):
- Meyer Children Hospital, Florence, Tuscany, Italy